CLINICAL TRIAL: NCT04684004
Title: Blood Glucose Values at Hospital Admission and Clinical Outcomes in Patients With Takotsubo Syndrome: Hyperglycemia Effects on Heart Failure Events and Mortality at 24 Months of Follow-up
Brief Title: Hyperglycemia in Patients With Takotsubo Syndrome
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, researcher, University of Campania Luigi Vanvitelli
Other Study IDs: 02.12.20
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Takotsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Death Domain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TTC patients with hyperglycemia: These patients will be hospitalized for TTC acute event. These patients will be characterized by higher blood glucose values at admission, and so defined as hyperglycemics.
  Interventions: Other: To report number of HF events and deaths
- TTC patients with normoglycemia: These patients will be hospitalized for TTC acute event. These patients will be characterized by normal blood glucose values at admission, and so defined as normoglycemics.
  Interventions: Other: To report number of HF events and deaths

INTERVENTIONS:
Other: To report number of HF events and deaths — In these two cohorts of study authors will evaluate at 2 years of follow-up the number of HF events and of deaths.

SUMMARY:
Patients with Takotsubo cardiomiopathy (TTC) have over-inflammation and over-sympathetic tone. However, these conditions could cause higher rate of heart failure (HF) events and deaths at 2 years of follow-up. Conversely, hyperglycemia vs. normoglycemia could result in over expression of inflammatory markers and catecholamines thta could result in higher rate of HF and deaths at 2 years of follow-up in TTC patients.

ELIGIBILITY:
Inclusion Criteria:

* acute onset of a cardiovascular event, usually associated with substernal chest pain, initially regarded as STEMI/evolving coronary syndrome;
* cardiac biomarker modifications (creatine kinase-MB and troponin I);
* systolic dysfunction, predominantly characterized by akinesia/hypokinesia of the mid-to-distal portion of the left ventricle (LV) chamber, with hyper-contractile basal LV.

Exclusion Criteria:

* patients with previous previous myocardial infarction;
* patients with previous TTC event;
* patients affected by chronic kidney, liver, and cerebrovascular diseases.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be of patients with acute TTC event. The enrolled patients according to inclusion and exclusion criteria will be then divided in normoglycemics vs. hyperglycemics according to blood glucose values at hospital admission.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
The number of HF events | 12 months
  To evaluate the number of HF events by clinical visits, telephonic interviews and hospital discharge schedules.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paolisso P, Bergamaschi L, Rambaldi P, Gatta G, Foa A, Angeli F, Fabrizio M, Casella G, Barbieri M, Galie N, Marfella R, Pizzi C, Sardu C. Impact of Admission Hyperglycemia on Heart Failure Events and Mortality in Patients With Takotsubo Syndrome at Long-term Follow-up: Data From HIGH-GLUCOTAKO Investigators. Diabetes Care. 2021 Sep;44(9):2158-2161. doi: 10.2337/dc21-0433. Epub 2021 Jun 29. PMID 34187841